CLINICAL TRIAL: NCT03828279
Title: The Global Registry on Hereditary Angioedema Type I and II
Brief Title: Global Registry to Gather Data on Natural History of Patients With Hereditary Angioedema Type I and II
Acronym: HGR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HAE Global Registry Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: HAERegistry
Record Dates: First submitted 2019-01-23; First posted 2019-02-04 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Hereditary Angioedema Type I and II
Keywords: angioedema; disease registry; C1 inhibitor; anti bradykinin treatments
MeSH Terms: conditions — Hereditary Angioedema Types I and II; Angioedema; Angioedemas, Hereditary | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Sodium Citrate samples are collected form patients for testing plasma levels of C1 inhibitor antigen and function and C4 antigen. Cells are collected for DNA extraction and detection of mutations in SERPING1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hereditary angioedema type I: Patients were diagnosed as C1 inhibitor HAE type I when functional and antigenic C1 inhibitor were ≤ 50% of normal
  Interventions: Diagnostic Test: functional and antigenic C1 inhibitor
- hereditary angioedema type II: Patients were diagnosed as type II when functional C1 inhibitor was ≤50% and antigenic was >50% of normal
  Interventions: Diagnostic Test: functional and antigenic C1 inhibitor

INTERVENTIONS:
Diagnostic Test: functional and antigenic C1 inhibitor — Diagnosis of HAE is based on personal and/or family history of angioedema and on C1 inhibitor functional or antigenic plasma levels ≤50% of normal.
  Other Names: genetic analysis

SUMMARY:
The objective of this international hereditary angioedema (HAE) register is to collect homogeneous clinical and laboratory data on patients with HAE type I and II gathering better information on the natural course of the disease and detecting therapeutic options to manage it.

DETAILED DESCRIPTION:
It is an international multicenter disease registry, the principal investigator at each center is responsible for competent ethic committee/institutional review board approval and for identifying co-investigators, who collect patients' informed consent and insert patients' data. Participating patients own their data. Upon acceptance of the informed consent, the treating physician transfers data of the case report form (CRF) to a specifically designed electronic support (eCRF) and the patients enter data on attacks. Physicians at center fill-in the eCRF with data for demography, diagnosis, prophylaxis and associated diseases. Plasma levels of C1 inhibitor antigen and function and of C4 antigen document laboratory diagnostic criteria. Each patient has a national identifier code. Patients fill-in attack reports that encompass duration, severity and treatment of each angioedema episode. C1 inhibitor coding gene (SERPING1) genotype is entered according to the last Hugo nomenclature. Yearly update of information is recommended, patients with follow up above two years are moved in a separate area and excluded from analysis. Each patient prospectively fills data on attacks. On a specific informed consent, the patient can agree on storing biological material (plasma and nucleic acids) for research purposes.

The data processor is an innovative start-up (Cloud-R s.r.l. Milan, Italy) that manages all data according to a specific contract and in compliance with current regulation on sensitive data security and processing. The Registry, delivered in the mode of Registry-as-a-Service (RaaS), is designed following General Data Protection Regulation (GDPR) guidelines, and issues regular software and infrastructure enhancements as a part of the normal operational mode. The system generates statistics of aggregated anonymized data following the participating centers' hierarchy levels and Global Registry governance rules. Patients supply data on attacks either on paper support or using a Web form or a mobile application. These data will flow into a staging area for physician validation before being considered valid for statistics. For each entry the system updates in real-time all the statistics and dashboards. The platform has configurable functionalities to support data quality management. It provides data format validation, integration to external qualified libraries, alerts, dashboards, automatic index calculations, advanced filters and queries, data change log. This open architecture, allows integration of the system, via standard API's, to external or sub-registries, registries, biobanks and clinical bioinformatics tools, i.e. for specific trial studies leveraging a specific cluster of patients already present in the Global Registry.

An independent non-profit foundation (HGRF) made of representatives of patients' associations is in charge for funding and delegates all the management to the HAE Global Registry Board (HGRB). The HGRB is in charge for operational, assisted by the HAE Global Registry Scientific Committee (HGRSC) for topics of competence. No registry member, center, group or board can access the entire set of data. All registry members, as single or group, can propose studies based on aggregated data by addressing the request to the HGRSC. Analysis and studies of data at local centers can occur at any time. Members of HGRB and HGRSC are elected to be representative of different cultural and geographic backgrounds. Their offices have a two-year term with no more than one consecutive renewal. Angioedema centers can join the Registry upon request to the HGRB . The registry quality control system periodically checks Registry entries and compliance of eCRF with the source data. For each information, the system will grant traceability of time and author.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with HAE type I and II with signed informed consent
* laboratory diagnostic criteria documenting plasma levels of C1 inhibitor antigen and function and of C4 antigen

Exclusion Criteria:

* patients without HAE type I and II
* patients without documented laboratory diagnostic criteria
* patients not capable to give informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with HAE type I and II and followed by a referral center for angioedema
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of angioedema events | Through study completion, an average of 5 years
  Number of angioedema events
Time of angioedema events | Through study completion, an average of 5 years
  Time in hours of presence of angioedema symptoms
Severity of angioedema events | through study completion, an average of 5 years
  Number of severe, moderate, mild angioedema symptoms based on a three point scale patient reported outcome

SECONDARY OUTCOMES:
Comorbidities | Through study completion , an average of 5 years
  Number and type of comorbidities recorded according to the International Classification of Diseases 9 codes
Treatment-Emergent comorbidities | Through study completion , an average of 5 years
  Incidence of comorbidities emerging in patients exposed to specific treatments
Treatment efficacy | Through study completion , an average of 5 years
  Hours of presence of angioedema symptoms during specific long term prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: marco cicardi, MD, Principal Investigator — HAE Global Registry Foundation
Locations (1):
- ASST FBF Sacco, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
All registry members, as single or group, can propose studies based on aggregated anonymized data by addressing the request to the HAE Global Registry Scientific Committee (HGRSC)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: entire study period
Access Criteria: to be a member of the HAERegistry and have the approval of the HGRSC to analyze data